CLINICAL TRIAL: NCT00072904
Title: Diabetes Therapy to Improve BMI and Lung Function in CF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Cystic Fibrosis Foundation (Other); Novo Nordisk A/S (Industry)
Responsible Party: Antoinette Moran, University Of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 58356DK (completed); NCT00177151 (obsolete NCT alias)
Record Dates: First submitted 2003-11-12; First posted 2003-11-14 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Cystic Fibrosis; Diabetes Mellitus
Keywords: Cystic Fibrosis Related Diabetes; Diabetes without Fasting Hyperglycemia
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus | interventions — repaglinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- III (Placebo Comparator): Placebo take half tab with meals tid
  Interventions: Drug: Insulin Asparte; Drug: Repaglinide

INTERVENTIONS:
Drug: Insulin Asparte — Insulin asparte given 0.5 units per carb per meal
Drug: Repaglinide — 0.5mg tab with meals tid

SUMMARY:
To recruit 150 adult patients with cystic fibrosis related diabetes (CFRD) without fasting hyperglycemia for a multi-center, twelve month, placebo-controlled intervention trial testing the ability of insulin or repaglinide to improve body mass index (BMI) and stabilize pulmonary function in cystic fibrosis (CF).

DETAILED DESCRIPTION:
The primary objective of this research is to determine whether treatment with either insulin or an oral diabetes agent that increases endogenous insulin secretion will improve BMI and pulmonary function in cystic fibrosis patients who have diabetes without fasting hyperglycemia.

ELIGIBILITY:
* Diabetic glucose pattern by oral glucose tolerance test (OGTT) of >200 at 120 min. (stable and healthy at time of OGTT)
* Fasting glucose levels <126.
* Weight stable within 5% in previous 3 months.
* Free from illness for two months.
* Male and female 16 and older, who are done growing
* Willing to come in for visits every 3 months.
* Patients receiving infrequent short bursts of systemic glucocorticoids may be considered for the study inclusion if: a. they have not received systemic glucocorticoids steroids for at least one month, b. they did not receive the steroids for more than 14 consecutive days or 28 days total in six months

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2001-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this research is to determine whether treatment with either insulin or an oral diabetes agent that increases endogenous insulin secretion will improve BMI and pulmonary function in cystic fibrosis patients who have diabetes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Moran, MD, Principal Investigator — University of Minnesota
Locations (7):
- United States (6):
  - Stanford University, Palo Alto, California
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Moran A, Pekow P, Grover P, Zorn M, Slovis B, Pilewski J, Tullis E, Liou TG, Allen H; Cystic Fibrosis Related Diabetes Therapy Study Group. Insulin therapy to improve BMI in cystic fibrosis-related diabetes without fasting hyperglycemia: results of the cystic fibrosis related diabetes therapy trial. Diabetes Care. 2009 Oct;32(10):1783-8. doi: 10.2337/dc09-0585. Epub 2009 Jul 10. PMID 19592632